CLINICAL TRIAL: NCT03975673
Title: Kinematic vs Mechanical Alignment Technique for Primary Total Hip Replacement in Patient With Hip Arthritis: a Prospective Comparative Non Randomised Study
Brief Title: Patient-Specific Techniques for Hip Replacement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre de l'arthrose, Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PST-HR
Record Dates: First submitted 2019-05-29; First posted 2019-06-05 (Actual); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Hip Arthritis; Hip Arthropathy
Keywords: hip arthroplasty; spine hip relation
MeSH Terms: interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Intervention Model Description: Prospective two-arms consecutive patients study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Total Hip Replacement (cTHR ) (Active Comparator): Osteoarthritic patient undergoing the conventional technique
  * medializing the hip center of rotation
  * obtain a standing acetabular cup position fitting the Lewinneck recommendations (inclination 40°±10°, version 15°±10°)
  Interventions: Procedure: hip replacement
- Kinematically Aligned Total Hip Replacement (KATHR ) (Experimental): Osteoarthritic patient undergoing the kinematically aligned technique
  * restoring the acetabular center of rotation
  * restoring the constitutional acetabular anteversion by using the transverse acetabular ligament (TAL) as a reference landmark.
  * making personalized choice for the hip component design
  * considering additional spine surgery based on the assessment of the individual spine-hip relation.
  Interventions: Procedure: hip replacement

INTERVENTIONS:
Procedure: hip replacement — Osteoarthritic patient undergoing the conventional technique or the kinematically aligned technique

SUMMARY:
Background

* In the 19th century, Sir John Charnley successfully introduced total joint replacements for hips. In order to prevent implant fixation failure and accelerated polyethylene wear, it was initially recommended that implants were systematically positioned in a "biomechanically-friendly" way, which disregarded most of the individual anatomy (medialized acetabular cup, systematized cup version and inclination, etc.)
* While those initial surgical techniques made popular and clinically successful total joint replacements, many complications (aseptic loosening, pain, excessive wear) have remained and mainly the persistence of frequent instability after THA. In response to those complications, many improvements were developed in the area of joint replacement over the last few decades, with one the most recent dating from 2017 and being the development of a surgical technique Rationale
* The kinematic alignment (KA) technique for total hip arthroplasty (THA) aims at restoring the acetabular center of rotation and as much as possible the constitutional acetabular anteversion by using the transverse acetabular ligament (TAL) as a reference landmark. Also, the technique aims (1) at making personalized choice for the hip component design, (2) at defining the cup positioning, and (3) at sometimes considering additional spine surgery based on the assessment of the individual spine-hip relation.
* KA techniques for hip replacements are relatively new, likely to become popular over time, and their true value remains to be determined.

DETAILED DESCRIPTION:
* Objective: Evaluation of the kinematic alignment technique for hip prostheses in patient with hip osteoarthritis
* Hypothesis: the consideration of hip pathoanatomy and lumbo-pelvic kinematic disorder when planning a hip replacement is likely to decrease the risk of prosthetic dislocation and improve patient function and satisfaction

ELIGIBILITY:
Inclusion Criteria:

* Osteoarthritic hip patients eligible for primary total hip arthroplasty (THR).
* > 18 years-old with no upper age limit
* Affiliated to a social security scheme

Exclusion Criteria:

* Pregnant or lactating women or in age to procreate without contraceptive treatment
* History of mental illness or neurological deficit or adults lacking capacity to consent for themselves
* Prisoners or young offenders
* Persons who might not adequately understand verbal explanations or written information given in French, or who have special communication needs
* Subjects having been or being frequently x-ray examination
* Heart failure with risk of exercise angina or comorbidity(ies) significantly affecting patient function
* Any participants who are involved in current research or have recently been involved in any research prior to recruitment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 460 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2020-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Dislocation rate | Occurrence within the first year after primary total hip replacement
  The rates of occurrence of hip dislocation (treated in the hospital or in an outpatient setting).

SECONDARY OUTCOMES:
EuroQualityOfLife 5 dimension index (EQ5D) | Preoperative, postoperative 6 months and 12 months . assessment for all parameters.
  EQ5D is a generic QoL scale from -0.6 to 1
Oxford hip score (OHS) | Preoperative, postoperative 6 months and 12 months . assessment for all parameters.
  OHS is a rate of hip function from 0 to 48
satisfaction visual analogic scale (VAS) | Preoperative, postoperative 6 months and 12 months . assessment for all parameters.
  satisfaction is a VAS score from 0 to 100
Implant positioning parameter | Preoperative, postoperative 6 months and 12 months . assessment for all parameters.
  Implant positioning parameters (inclination, version, offset) are computed on post-operative X rays acquisition.

CONTACTS AND LOCATIONS:
Overall Officials: Cedric Maillot, Principal Investigator — centre de l'arthrose
Locations (1):
- Université de Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No